CLINICAL TRIAL: NCT05279794
Title: Efficacy of Two Types of Non-invasive Erector Spinae Muscle Taut Band Therapy in University Students With Low Back Pain: A Randomized Clinical Trial
Brief Title: Efficacy of Two Types of Non-invasive Erector Spinae Muscle Taut Band Therapy in University Students With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Martínez Fuentes, Study Director, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE012207
Record Dates: First submitted 2022-02-07; First posted 2022-03-15 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Low Back Pain; Trigger Point Pain, Myofascial
Keywords: Physiotherapy; Rehabilitation; Treatment; Active Trigger Point
MeSH Terms: conditions — Low Back Pain; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jones Group (Strain Counterstrain) (Experimental): Jones Group consist in 90 seconds in a ralease positioning of no pain in muscle acortation
  Interventions: Other: Jones Group (Strain Counterstrain)
- Myofascial Induction Group (Active Comparator): Myofascial Induction Group consist in 15 minutes of superficial and deep lumbar fascia maneuvers
  Interventions: Other: Myofascial Induction Group
- Placebo Group (Placebo Comparator): Placebo Group only have to mantain no pain positioning for 3 minutes
  Interventions: Other: Placebo Group

INTERVENTIONS:
Other: Jones Group (Strain Counterstrain) — No pain positioning technique with diaphragmatic breathing
  Arms: Jones Group (Strain Counterstrain)
Other: Myofascial Induction Group — Myofascial Induction technique on the lumbar fascia
  Arms: Myofascial Induction Group
Other: Placebo Group — No pain positioning of participants
  Arms: Placebo Group

SUMMARY:
Non-specific low back pain can be caused by the presence of active trigger points in the muscles of the lumbopelvic region. Trigger points are defined as hypersensitive points within a taut band of a musculoskeletal system that cause pain during contraction, stretching, or stimulation of said muscle. If these points are active, they can trigger referred pain, local tenderness, and vegetative responses. There is scientific evidence of the improvement of the treatment of these points through non-invasive manual techniques. The objective of this study will be to determine the effect of Strain Counterstrain and Myofascial Induction techniques in subjects with low back pain secondary to the presence of active trigger points in the lumbopelvic region. Hyperexcitable myofascial trigger points located within a taut band of skeletal muscle or fascia cause referred pain, local tenderness, and autonomic changes. The scientific data refer to an immediate improvement in the symptoms of these active points treated with manual therapy. Based on these factors, the objective of the study is to determine the effect of the combined therapy of the Strain Counterstrain technique and Myofascial Induction in participants with the presence of an active trigger point in the erector spinae muscle.

DETAILED DESCRIPTION:
The treatment will last a total of 15 minutes accompanied by a baseline assessment and after 10 minutes of the intervention in 2 experimental groups and a placebo group, of no-pain positioning. In addition to basic indices and scales of low back pain and disability caused by low back pain, it is intended to measure flexibility, range of motion, proprioception and cognition through software with sensors of the latest technology when representing reliable results in differences between techniques.

ELIGIBILITY:
Inclusion Criteria:

* Presence of low back pain
* Presence of active trigger point in the erector spinae as described by Lawrence H. Jones

Exclusion Criteria:

* Participants who present dizziness, vertigo;
* Previous or scheduled surgeries in the lumbar spine and/or lower extremities;
* Suspicion of serious fractures or pathologies (tumor, inflammation, infection, rheumatological disorder, systemic disease, presence of fever);
* Diagnosis of radiculopathy or neuropathy;
* Structural deformity in the spine; spondyloarthropathy, disabling pain and physical disability;
* Use of pain relievers or anti-inflammatory drugs in the last 48 hours;
* Neurological or psychiatric disorder;
* Presence or suspicion of pregnancy

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 20 minutes
  Measured with Numeric Rating Scale wich consist in measure pain intensity with a score of 0-10
Pression algometer | 20 minutes
  Measures pressure pain thresholds

SECONDARY OUTCOMES:
Spinal test | 20 minutes
  Measured with Baiobit Software. The range of movement will be measured in grades as per: flexion/extension; right/left rotation; and right/left inclination
Countermovement jump test | 20 minutes
  Measured with Baiobit software counter movement jump test wich consist a velocity, height and accuracy evaluation of a vertical jump

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Murcia, Murcia, Spain